CLINICAL TRIAL: NCT02475057
Title: A Pilot Study on Endothelial Function and Cardiovascular Biomarkers in Prostate Cancer (PCa) Patients, With Pre-existing Cardiovascular Disease, Treated With Degarelix vs. Luteinizing Hormone-Releasing Hormone (LHRH) Agonists
Brief Title: Endothelial Function in Prostate Cancer Patients on Degarelix vs. Luteinizing Hormone-Releasing Hormone Agonists
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0102-15-RMC
Record Dates: First submitted 2015-06-08; First posted 2015-06-18 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Prostatic Neoplasms; Cardiovascular Diseases
Keywords: Prostate Cancer; Cardiovascular disease; Degarelix
MeSH Terms: conditions — Prostatic Neoplasms; Cardiovascular Diseases | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Degarelix (LHRH antagonist) (Experimental): Degarelix (LHRH antagonist) EndoPAT2000
  Interventions: Drug: Degarelix (LHRH antagonist); Device: EndoPAT2000
- LHRH agonist (Active Comparator): LHRH agonist at the discretion of the treating Urologist/Oncologist EndoPAT2000
  Interventions: Drug: LHRH agonist; Device: EndoPAT2000

INTERVENTIONS:
Drug: Degarelix (LHRH antagonist) — Two initial loading doses of 120mg Degarelix for 1 month followed by 80mg monthly for eleven additional months.
  Other Names: Firmagon
  Arms: Degarelix (LHRH antagonist)
Drug: LHRH agonist — LHRH agonist at the discretion of the treating Urologist/Oncologist for 1 year.
  Other Names: Luteinizing hormone-releasing hormone agonist
  Arms: LHRH agonist
Device: EndoPAT2000 — Peripheral arterial plethysmography using an EndoPAT2000 device
  Other Names: Peripheral arterial plethysmography

SUMMARY:
The purpose of this study is to test whether Degarelix is associated with less endothelial dysfunction (an intermediate in the development of cardiac disease) and cardiovascular biomarkers compared to LHRH agonists.

DETAILED DESCRIPTION:
This is a national multicenter randomized open-label superiority study of the use of Degarelix compared to LHRH agonists among men with advanced prostate cancer and pre-existing cardiovascular disease. Patients will be stratified based on baseline endothelial function and presence prostate cancer metastasis.

Study population: Subjects with pre-existing cardiovascular disease with locally advanced or metastatic prostate cancer and scheduled to start Androgen Deprivation Therapy (ADT). Patients already on ADT will be excluded. subjects will receive either two initial loading doses of 120mg Degarelix for 1 month followed by 80mg monthly for eleven additional months or an LHRH agonist at the discretion of the treating Urologist/Oncologist for 1 year. Follow-up visits will occur every 3 months. A blood sample for Prostate-specific antigen (PSA), cardiac biomarkers and rectal examination will be performed each visit. At baseline 6 and 12 months EndoPAT2000 measurements will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with locally advanced or metastatic prostate cancer or high-risk prostate cancer.
* Scheduled to start ADT for a period of at least one year.
* Subject has a history of one or more of the following:

  1. Myocardial infarction
  2. Ischaemic or Haemorrhagic cerebrovascular conditions
  3. Arterial embolic and thrombotic events,
  4. Ischaemic heart disease
  5. Prior coronary artery or iliofemoral artery revascularization (percutaneous or surgical procedures)
  6. Peripheral vascular disease (e.g. significant stenosis (ABPI<0.9), claudication, prior vascular surgery/intervention)
* Life expectancy of over 12 months.
* WHO performance status of 0-2
* Subject is able and has agreed to sign a consent form.

Exclusion Criteria:

* Prior use of ADT. However, prior use of anti-androgens such as Casodex, Chimax, Drogenil, and Cyprostat will be allowed.
* Prior use of dutasteride/finasteride in past 6 months
* Known allergic reaction to Degarelix.
* Any psychological, familial, sociological or geographical situation potentially hampering compliance with the study protocol and follow-up schedule.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in Reactive Hyperemia Index from baseline to twelve months | Baseline, and twelve months
  the Reactive Hyperemia Index is a measure of endothelial function. It will be measured using the EndoPAT2000

SECONDARY OUTCOMES:
Change in High sensitivity troponin (hsTn) value | Baseline, and after three, six and twelve months of treatment initiation
  High sensitivity troponin (hsTn) is a biomarker for acute myocardial injury
Change in C-reactive protein value | Baseline, and after three, six and twelve months of treatment initiation
  C-reactive protein is a biomarker for inflammation
Change in D-dimer value | Baseline, and after three, six and twelve months of treatment initiation
  D-dimer is a biomarker for coagulation system activation
Change in N-terminal pro-brain natriuretic peptide (NT-proBNP) value | Baseline, and after three, six and twelve months of treatment initiation
  N-terminal pro-brain natriuretic peptide (NT-proBNP) is a biomarker for myocardial strain

OTHER OUTCOMES:
Change in testosterone level | Baseline, and after three, six and twelve months of treatment initiation
Change in gonadotropins levels | Baseline, and after three, six and twelve months of treatment initiation
  LH
Change in PSA value | Baseline, and after three, six and twelve months of treatment initiation
  Prostate-specific antigen
Change in BMI | Baseline, and after three, six and twelve months of treatment initiation
  Body Mass Index
Change in Quality Of Life score | Baseline, and after three, six and twelve months of treatment initiation
  As assessed by the FACT-P quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Margel, MD, PhD, Principal Investigator — Rabin Medical Center
Locations (2):
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976